CLINICAL TRIAL: NCT06450743
Title: Age-matched Reference Values for Circulating Natural Killer t (NKT)-Like Cells
Brief Title: Age-matched Reference Values for Circulating Natural Killer T-like Cells
Acronym: NKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0014476
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Lymphocytes; NKT-like cells; Reference Values

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Derivation Cohort (Other): Adult and pediatric patients who have routinely performed the lymphocyte immunophenotyping test, including also the enumeration of NKT-like cells, to exclude an immunological impairment during the period from May 2019 to March 2020 (for adults) and from May 2019 to August 2021 (for pediatric patients).
  Interventions: Diagnostic Test: Lymphocyte Immunophenotyping Test
- Validation Cohort (Other): Healthy adult blood donors in order to validate the obtained results.
  Interventions: Diagnostic Test: Lymphocyte Immunophenotyping Test

INTERVENTIONS:
Diagnostic Test: Lymphocyte Immunophenotyping Test — Absolute enumeration of peripheral blood lymphocyte subpopulations

SUMMARY:
Few data are so far available regarding the adult normal values of circulating NKT-like cell concentration, and none for the pediatric population. The primary objective of this study is to determine the reference values for NKT-like cells in pediatric and adult patients (derivation cohort). The secondary objective is to validate the results obtained from the adult derivation cohort with those obtained from an adult validation cohort, consisting of a group of healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy blood donor
* without acute or chronic pathological conditions
* matched for sex and age with the retrospective adult derivation cohort

Exclusion Criteria:

* a history of immunological or hematological diseases, immunosuppressive or immunostimulant therapies, or ongoing infections
* one of the lymphocyte subpopulations tested out of range
* undergoing surgery or dentistry intervention in the past two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
NKT-like cells reference values determination (absolute number and percentage) from the derivation cohort | 2 months
  Retrospective analysis of NKT-like cell counts from the lymphocyte immunophenotyping test performed on adult (>16 years) and pediatric outpatients divided in narrow age ranges (0-15 months, 15-24 months, 2-5 years, 5-10 years, 10-16 years) to obtain reference values.

SECONDARY OUTCOMES:
NKT-like cells reference values validation (absolute number and percentage) using healthy blood donors (>16 years) | 1 month
  Analysis of NKT-like cell counts from the lymphocyte immunophenotyping test on healthy adult blood donors and comparison with those obtained from adult patients of derivation cohort to verify that will not statistically differ.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Trombetta, BSc, Principal Investigator — Flow Cytometry Laboratory, Clinical Pathology
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No